CLINICAL TRIAL: NCT06503419
Title: Caregiver Burden, Quality of Life, Family Function and Family Resilience Among Caregivers of Children With Medical Complexity: A Mixed Methods Convergent Parallel Design
Brief Title: Caregiver Burden, Quality of Life, Family Function and Family Resilience Among Caregivers of Children With Medical Complexity.
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202406005RINE
Record Dates: First submitted 2024-07-01; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Caregiver Burden; Quality of Life; Family Function; Family Resilience
Keywords: Children with medical complexity; caregiver burden; quality of life; family functioning; family resilience
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
The purpose of this study is to employ a mixed methods research approach combining quantitative and qualitative methods to thoroughly understand the relationships among caregiver burden, quality of life, family functioning, and family resilience of children with medical complexity (CMC). The study aims to explore the individual and social factors influencing these variables and investigate the factors impacting caregiver burden, quality of life, family functioning, and family resilience of CMC caregivers. Finally, an integrative analytical framework will be proposed. The study seeks to provide guidance and recommendations for social support for caregivers of children with medical complexity in caregiving practices, aiming to promote the development of relevant policies and services.

DETAILED DESCRIPTION:
This study employs a convergent parallel mixed methods design. The quantitative part involves a questionnaire survey using purposive and snowball sampling methods, inviting 400 caregivers of children with medical complexity (CMC) to participate. Stratified sampling is then applied, with 62 samples selected per age group (1-5 years, 6-10 years, 11-15 years, 16-20 years), resulting in a total of 248 valid samples. The aim is to measure the correlations among caregiver burden, quality of life, family functioning, and family resilience. For the qualitative research, purposive and snowball sampling methods are also used to recruit 10 caregivers of CMC from different age groups who meet the inclusion criteria and agree to participate. These caregivers undergo semi-structured in-depth interviews, with interview content recorded to gain deeper insights into their experiences and feelings regarding caregiver burden, quality of life, family functioning, and family resilience. The study instruments include validated tools such as the Caregiver Burden Inventory (CBI), SF-12 Health Survey for quality of life, the APGAR Family Functioning Scale, and a Chinese version of the Family Resilience Scale. Qualitative data are collected through semi-structured interviews. Data analysis involves descriptive statistics, analysis of variance (ANOVA), and multiple linear regression models using IBM SPSS Statistics 27 for quantitative data. Qualitative data are analyzed using textual and thematic analysis methods, supported by NVivo qualitative analysis software. Finally, data triangulation is employed to integrate and compare quantitative and qualitative findings, leading to conclusions and recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Must be the primary caregiver of a child with medical complexity, providing care for at least 12 months.
2. Aged 20 years or older.
3. Must be a cohabiting family member of the child and have a biological relationship with the child.
4. Willing to participate in the study.
5. The child with medical complexity being cared for by the participant is between the ages of 1 and 20, diagnosed by a physician with a chronic illness or disability. The child requires the use of medical equipment or devices at home, including respiratory support equipment such as tracheostomy care supplies, artificial ventilation masks, mechanical ventilators (respirators), oxygen concentrators and tanks, suction machines, and percussion vests; nutritional and medication devices such as gastric tubes (nasogastric or percutaneous gastrostomy tubes), enteral feeding pumps, and intravenous catheters; mobility aids including wheelchairs, walkers, and rehabilitation assistive devices; monitoring equipment such as electrocardiogram (ECG) monitors, blood pressure monitors, thermometers, and pulse oximeters; and other medical equipment such as urinary bags and catheters, and pain management pumps (e.g., PCA). Additionally, due to their condition, the child receives regular medical examinations or treatments.

Note: Inclusion criteria are the same for both quantitative and qualitative studies.

Exclusion Criteria:

1. Diagnosed with a mental illness by a physician.
2. Assessed by the researcher as lacking the reading and comprehension abilities necessary to complete the study.

Note: Exclusion criteria are the same for both quantitative and qualitative studies.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises primary caregivers of children with medical complexity (CMC)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden Inventory (CBI) | Less than 1 hour.
  Scale: 0 to 96, with higher scores indicating greater caregiver burden. Description: This measure will assess the time dependence, developmental, physical, social, and emotional burdens experienced by caregivers of children with medical complexity.
Quality of Life [Short Form Health Survey (SF-12)] | Less than 1 hour.
  Scale: 0 to 100 for each domain, with higher scores indicating better quality of life.
  Description: This measure will evaluate the physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health of caregivers.
Family Function (Family APGAR) | Less than 1 hour.
  Scale: 0 to 10, with higher scores indicating better family function. Description: This measure will assess family adaptability, partnership, growth, affection, and resolve.
Family Resilience Scale | Less than 1 hour.
  Scale: 31 to 155, with higher scores indicating greater family resilience. Description: This measure will evaluate the belief systems, organizational patterns, and communication processes of families dealing with children with medical complexity.
Qualitative Understanding of Caregiver Experiences by Semi-structured Interviews | About 1 hour.
  This measure will complement the quantitative data by providing in-depth insights into the personal experiences, challenges, coping strategies, and perspectives of caregivers of children with medical complexity. Thematic analysis will be conducted on the qualitative data to identify key themes and factors influencing caregiver burden, quality of life, family function, and family resilience.Description: This measure will complement the quantitative data by providing in-depth insights into the personal experiences, challenges, coping strategies, and perspectives of caregivers of children with medical complexity.

CONTACTS AND LOCATIONS:
Overall Officials: ChingWen Cheng, MD, Study Chair — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No